CLINICAL TRIAL: NCT07004855
Title: Tai Po Hidden Carers Support and Home-Based Respite Project
Acronym: VRDCFIn-home2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Vivian W.Q. Lou, Director, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EA250321
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Caregiver Wellbeing
Keywords: caregiver; respite
MeSH Terms: interventions — Crew Resource Management, Healthcare

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Caregiver - Low level (Experimental): Caregivers in low level will receive case follow-up service from social workers
  Interventions: Other: Case follow-up
- Caregiver - Mild level (Experimental): Caregivers in mild level will receive regular phone check-in and on-demand services provided by volunteers
  Interventions: Other: Phone Check-in
- Caregivers - Moderate level (Experimental): Caregivers in moderate level will receive 30 hours of respite service within 6 months
  Interventions: Other: 30 hr Respite Service
- Caregiver - High level (Experimental): Caregivers in high level will receive crisis management and counselling from social workers and professionals.
  Interventions: Other: Crisis management

INTERVENTIONS:
Other: 30 hr Respite Service — Caregivers will be provided with 30 hours of respite service within 6 months. Trained substitute caregivers will provide in-home elderly-sitting service.
  Arms: Caregivers - Moderate level
Other: Case follow-up — Case follow-up service provided by social workers. Social workers will call the caregiver regularly to see if situation changes.
  Arms: Caregiver - Low level
Other: Crisis management — Crisis management and councelling provided by social workers and professionals.
  Arms: Caregiver - High level
Other: Phone Check-in — Regular phone check-in and on-demand services (e.g., escort to hospital) provided by volunteers.
  Arms: Caregiver - Mild level

SUMMARY:
The primary objective of this study is to identify and support hidden caregivers of older adults. Caregivers are assessed before the intervention on their mental well-being and social connectedness. Caregivers are triaged into four levels: low, mild, moderate and high. They will receive different types of services (intervention) accordingly. At the end of the service period (or 6-months after the baseline), caregivers and care recipients will complete the assessment again to measure the changes of the primary outcomes.

DETAILED DESCRIPTION:
"All participants will provide informed consent at the time of enrolment. Both caregivers and their care recipients will complete an assessment. Caregivers are screened for their physical health, mental well-being, social engagement, and social connectedness. Care recipients are screened for their physical health and capacity in activities of daily living and instrumental activities of daily living.

Caregivers are triaged into four levels: low, mild, moderate and high. Caregivers in low level will receive case follow-up service, those in mild level will receive regular phone check-in, those in moderate level will receive a maximal of 30 hours of respite service within 6 month, and those in high level will receive professional counselling. At the end of the service period (or 6-months after the baseline), caregivers and care recipients will complete the assessment again to measure the changes of the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Provide ADL/IADL assistance to at least one older adult (aged 60+),
* Not currently using any types of respite service,
* Able to communicate in either Cantonese, English or Mandarin
* Voluntarily participate

Exclusion Criteria:

* The care recipient is not living in the community

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in score in caregiving needs on the Carer Needs Screening Tool (CNST-11) after the intervention | Baseline and Immediate after intervention
  The Carer Needs Screening Tool (CNST-11) is a self-developed tool that measures different aspects of caregiving needs over the past 1 week period. It is a 11-item scale, with 8 items that determines the overall needs level and the others for four aspects of needs: physical health, mental health, social support and care needs. Possible score is from 8 to 32 with lower score indicates lower caregivers' needs.
  Change in score = Immediate after intervention - baseline
Change from baseline in score in social support on MOS Social Support Survey after the intervention | Baseline and Immediate after intervention
  The MOS Social Support Survey (MOSSSS) is a widely used tool that consists of 6 questions designed to measure the amount of support one needs. The total score ranges from 6 to 30, with higher scores indicating more support received.
  Change in score = Immediate after intervention - baseline
Change from baseline in score in the severity and disturbance of symptoms of care recipient on Neuropsychiatric Inventory after the intervention | Baseline and Immediate after intervention
  The Neuropsychiatric Inventory measures the severity and disturbance to caregiver of 13 common symtoms (e.g., dellusion, sleeping problem) of the care recipient. Severity is rated from 0 to 3, with 0 indicates no symptom and 3 indicates severe problem. Disturbance to caregiver is rated from 0 to 5, with 0 being not affected at all and 5 being extremely affected. The higher score in both subscales indicate worse problem.
  Change in score = Immediate after intervention - baseline
Change from baseline in score in social connectedness on Social Connectedness Scale after the intervention | Baseline and Immediate after intervention
  The Social Connectedness Scale consists of 6 items that measures how closely one feel that they are connected to the community. The total score on the scale can range from 8 to 48, with higher scores indicating a higher level of connectedness.
  Change in score = Immediate after intervention - baseline
Change from baseline in score in the view on gender role on Gender Role Attitude Scale after the intervention | Baseline and Immediate after intervention
  The Gender Role Attitude Scale consists of 3 items that measure the view on traditional gender role. The total score range from 3 to 15, with lower score indicate more traditional value.
  Change in score = Immediate after intervention - baseline
Change in score from baseline in quality of life measured by EQ-5D-5L after intervention | Baseline and Immediate after intervention
  The EQ-5D-5L is a standardized instrument used to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The responses are converted into a single index value representing overall health status using Hong Kong's normative value. The primary outcome measure in this study is the change in EQ-5D-5L index scores from baseline to post-intervention/follow-up assessments. 1 equals to perfect health and more negative numbers indicates worse health. Change in health index = Immediate after intervention - baseline
Changes in score from baseline in perception of caregiving measured by Positive Aspect of Caregiving scale after intervention | Baseline and Immediate after intervention
  The Positive Aspect of Caregiving scale is a 11-item scale that measures how the caregiver perceive caregiving experience, specifically in a positive aspect (e.g., caregiving makes me feel useful). It is rated in a 5-point Likert scale from "very disagree" to "very agree", with potential score from 0 to 44. A higher score indicates caregiving perceiving it in a more positive way.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Informed consent form and anonymous data will be uploaded to HKU Data Repository under embargo protection.
Supporting Information: ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Informed consent form and anonymous data will be uploaded to HKU Data Repository under embargo protection.